CLINICAL TRIAL: NCT05499650
Title: The Effects of Exercise on Quality of Life and Fluid Dynamics in Patients With Aortic Dissection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No sufficient eligible participants identified.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Areck Ucuzian, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00099260
Record Dates: First submitted 2022-08-03; First posted 2022-08-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Aortic Dissection
Keywords: Exercise; Fluid Dynamics; Quality of Life
MeSH Terms: conditions — Aortic Dissection; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Group (Experimental): Patients will be required to undergo an exercise program. Pre-intervention and post-intervention outcomes will be compared in each patient.
  Interventions: Behavioral: Supervised Exercise Regiment

INTERVENTIONS:
Behavioral: Supervised Exercise Regiment — Subjects will undergo supervised aerobic exercise. There will be a set goal mean energy expenditure of at least 1000 kcal/wk after a two-week ramp-up period. The protocol will include 30 minutes of moderate-intensity exercise with a treadmill and cycle ergometry, two times weekly. Strenuous resistance training and swimming will be withheld from this protocol due to the potential concerns for safety in exacerbating dissections. Heart rate and ratings of perceived exertion will be quantified during the therapy with a standard set heart rate ad pulse pressure threshold for discontinuing exercise protocols.

SUMMARY:
Aerobic exercise and physical activity improve patient health in patients in a variety of aspects of life and disease. It also improves patients' mental well-being and quality of life. However, the safety of this physical activity and its potential benefits remain uncertain for patients after aortic dissection, a tear in the main blood vessel delivering blood to all of the body's organs.

The goal of this study is to facilitate the translation of pre-clinical findings by the Principal Investigator and published literature that demonstrates light to moderate exercise is safe and beneficial in patients with thoracic aortic dissection. This will be accomplished by using both imaging-based analyses of aortic wall responses to a 3- month exercise program, patient surveys of quality of life metrics, functional fitness assessments, and clinical outcomes.

DETAILED DESCRIPTION:
This is a pilot longitudinal study with the primary goal of validating preclinical results and demonstrating the safety and feasibility of moderate aerobic exercise in patients with aortic dissection. The study will enroll 5 patients with a history of aortic dissection >90 days from inciting event treated either operatively or non-operatively. Future studies will recruit a larger cohort of patients.

In addition to standard therapy, subjects will undergo supervised aerobic exercise, with a set goal mean energy expenditure of at least 1000 kcal/wk.

Based on the literature, and preliminary data, it is anticipated that exercise therapy initiated in conjunction with standard of care medical and surgical management of type B thoracic aortic dissection is safe and improves patient quality of life. Subjects will undergo supervised aerobic exercise. Baseline testing includes a CT with a standard protocol for high resolution imaging of the vasculature called a CT angiogram (CTA), cardiopulmonary exercise testing, maximal oxygen consumption (peak VO2) during a treadmill test, and arterio-venous differences, a quality-of-life questionnaire, and an assessment of activity at baseline with the 7- day activity recall questionnaire, this will be obtained between the clinic visit at which informed consent is obtained and initiation of the study. In addition to baseline testing, cardiopulmonary testing, a quality-of-life questionnaire, and an assessment of activity at baseline with the 7-day activity recall questionnaire will occur at 3 months. CTA will occur at baseline (if none exists within 30 days) and at 3 months. 3-month data will be compared with baseline data and analyzed by a paired T-test for continuous data. In addition to baseline testing cardiopulmonary testing, a quality-of-life questionnaire and an assessment of activity at baseline with the 7-day activity recall questionnaire will occur at 3 months, as well as a CTA. The 3-month data will be compared with baseline data and analyzed by a pair of T-tests for continuous data.

Patients will also receive standard therapy for the management of chronic aortic dissection. This includes adequate blood pressure control and heart rate control with beta-blockers or calcium-channel blockers. A standard therapy will allow the real-world practice of standard of care for the medical goals of maintenance of systolic blood pressure between 100-120 mm Hg. And heart rates with 60-80 beats per minute. Patients will be directed not to partake in strenuous resistance exercises such as weight-lifting, but will also not be given direction regarding the amount of activity they should adhere to on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 88
* History of aortic dissection > 90 Days from acute event
* Previous operative or non-operative management of aortic dissection
* Ability to undergo basic level of activity and exercise
* Able to consent
* Capable of basic communication and recall

Exclusion Criteria:

* History of surgically untreated Type A Dissection
* Patients within 90 days of acute dissection event
* Patients with unstable coronary artery disease
* Patients with severe cardiopulmonary disability (class III/IV heart failure and/or ejection fraction < 20%),
* Patients with malignant hypertension
* Patients with previous stroke with significant persistent motor deficit
* Patients with any orthopedic or podiatric conditions altering their ambulation status will be excluded.
* Patients with any other health reasons which preclude exercise tolerance such as morbid obesity (BMI > 39 kg/m2), severe hepatic dysfunction, critical aortic stenosis, or active pericarditis or myocarditis.
* Patients with allergies to iodinated contrast as would be used for CT scan surveillance.
* Patients who have significant barriers for reliable follow-up
* Patients with significant cognitive impairment, or who are unable to carry-out basic communication and recall.
* Patients belonging to vulnerable populations
* Patients with connective tissue disorders such as Marfan's syndrome, Ehlers-Danlos Type IV, or Loesz-Dietz syndrome
* Patients who are unable or unwilling to consent
* Age less than 18 or over 88.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Health related Quality of Life (HRQOL) scores | 3 months
  0-30 Unhealthy days, lower being better
Physical Activity Scale for the Elderly (PASE) scores | 3 months
  0-400, Higher being better

SECONDARY OUTCOMES:
Aortic Shear Stress | 3 months
  Pascal; CT-based Computation fluid dynamics will determine pre and post-exercise regimen change in aortic shear stress
Maximal oxygen consumption during Exercise (V02 Max) | 3 months
  A fitness measurement (higher number indicates higher fitness). This estimate uses the ratio of maximum heart rate (HRmax) to resting heart rate (HRrest) to predict V̇O2 max (mL/kg/min).
Number of aortic related hospitalization | 1 year
  Observational aortic related hospitalizations (admission requirement secondary to acute aortic pathology)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No